CLINICAL TRIAL: NCT02973282
Title: Diagnosing Respiratory Disease in Children Using Smartphone Recordings of Cough Sounds
Brief Title: Diagnosing Respiratory Disease in Children Using Cough Sounds
Acronym: SMARTCOUGH-C
Status: Completed | Type: Observational
Sponsor: ResApp Health Limited (Industry)
Collaborators: Massachusetts General Hospital (Other); The Cleveland Clinic (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 16001
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Pneumonia; Bronchiolitis; Asthma; Croup; Upper Respiratory Tract Infection; Lower Respiratory Tract Infection; Reactive Airway Disease
MeSH Terms: conditions — Pneumonia; Bronchiolitis; Asthma; Croup; Respiratory Tract Infections; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Recording of Infants and Children's Cough Sounds — Smartphone recordings of the cough sounds of infants and children presenting to a participating site with signs or symptoms of respiratory disease

SUMMARY:
The purpose of this prospective study is to evaluate the efficacy of the ResAppDx software application in diagnosis of pneumonia and other respiratory conditions (bronchiolitis, asthma/reactive airway disease, croup, upper or lower respiratory tract infections) in infants and children. Patient's cough sounds will be recorded using a smartphone and analysed using the ResAppDx software. The ResAppDx diagnosis will be compared to radiologic diagnosis and/or clinical diagnosis. The ResAppDx diagnosis will not be provided to the clinician or patient.

ELIGIBILITY:
Inclusion Criteria:

* Infant or child aged 29 days - 12 years
* Presenting to the study site with signs or symptoms of respiratory disease including cough, wheezing, stridor, chest in-drawing/retractions, difficulty breathing, fast breathing, abnormal lung sounds on exam, cyanosis/hypoxemia.
* Coughing spontaneously or able to cough voluntarily

Exclusion Criteria:

* Lack of a signed consent form from parent or legal guardian
* Lack of signed assent form for children aged 7 years or older who, in the opinion of the investigator, is able to provide assent based on their age, maturity or psychological state.
* Need for mechanical ventilatory support (including invasive, continuous positive airway pressure, or bilevel positive airway pressure) or high flow nasal cannula
* Any medical contraindication to voluntary cough, including (only enrolled if coughing spontaneously): severe respiratory distress, history of pneumothorax, eye/chest/abdominal surgery in past 3 months, hemoptysis in the past month, or too medically unstable to participate in study per treating clinician.
* Subject previously enrolled
* Tracheostomy present or tube placed

Ages: 29 Days to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with signs or symptoms of respiratory disease presenting to participating Emergency Departments, Urgent Care Clinics, Primary Care Clinics
Sampling Method: Non-Probability Sample
Enrollment: 1245 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of pneumonia | 6 months
  Positive percent agreement and negative percent agreement to diagnose and rule out pneumonia as compared with a radiologic diagnosis.
  Positive percent agreement and negative percent agreement to diagnose and rule out pneumonia as compared with a clinical diagnosis.

SECONDARY OUTCOMES:
Diagnosis of other childhood respiratory diseases | 6 months
  Positive percent agreement and negative percent agreement to diagnose and rule out: lower respiratory tract involvement, bronchiolitis, asthma/reactive airway disease, upper respiratory tract infection and/or croup, as compared with a clinical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Moschovis, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No